CLINICAL TRIAL: NCT07165158
Title: The Effect of Semaglutide on Osteoporotic Fractures in Patients With Type 2 Diabetes
Brief Title: The Effect of Semaglutide on Bone Health
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The First Affiliated Hospital of Xiamen University (Other)
Collaborators: Peking University First Hospital (Other); Shanghai Punan Hospital of Pudong New District (Other); Shanghai 6th People's Hospital (Other); Jinzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: KYLLPJ2025-033
Record Dates: First submitted 2025-09-01; First posted 2025-09-10 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-08

CONDITIONS: Osteoporosis; Osteoporosis Fracture; T2DM
Keywords: antidiabetic drug; osteoporosis fracture; T2DM
MeSH Terms: conditions — Osteoporosis; Osteoporotic Fractures | interventions — Metformin

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The intervention group (Experimental): In the intervention group, the participants will receive semaglutide combined with metformin treatment.
  Interventions: Drug: semaglutide combined with metformin
- The control group (No Intervention): In the control group, the participants will be treated with metformin alone (500mg each time, three times a day).

INTERVENTIONS:
Drug: semaglutide combined with metformin — The initial dose of semaglutide is 0.25 mg once weekly. After 4 weeks, the dose is adjusted to 0.5 mg once weekly. After another 4 weeks, the dose is adjusted to 1 mg once weekly. During the same period, they will take metformin (500mg each time, three times a day) for treatment. The treatment course is 12 months.
  Arms: The intervention group

SUMMARY:
Semaglutide has effects that include lowering blood sugar, reducing weight, and improving cardiovascular and renal outcomes, and it is now widely used in clinical practice. Given that weight loss is associated with bone loss, its effect on bone health has recently raised concerns. Therefore, the goal of this clinical trial is to learn the effect of semaglutide on bone mineral density and fractures in patients with type 2 diabetes.

The investigators will compare semaglutide combined with metformin to metformin alone to see if semaglutide treatment has effects on bone mineral density and bone turnover markers in patients with type 2 diabetes after 12 months.

The intervention group will receive semaglutide combined with metformin for 12 months, while the control group will receive metformin alone for the same duration. After 12 months of treatment, the investigators will compare the bone mineral density, fracture incidence, and levels of bone turnover markers between the two groups.

ELIGIBILITY:
Inclusion Criteria:

1. Type 2 diabetes (according to WHO diagnostic criteria),
2. Age range: 50 to ≦75 years,
3. Glycosylated hemoglobin (HbA1c): 6.5 to ≦9.0%,
4. Bone mineral density (lumbar spine, hip, or femoral neck) T-score < -1, or history of fragility fractures (hip, vertebral, distal forearm, or proximal humerus fractures) within three years before screening,
5. No use of antidiabetic medications in 8 weeks prior to enrollment (excluding metformin).

Exclusion Criteria:

1. Bone mineral density (lumbar spine, hip, or femoral neck) T-score < -2.5,
2. History of secondary osteoporosis,
3. Serious liver dysfunction or chronic kidney disease (aspartate aminotransferase (AST) or alanine transaminase (ALT) > 2.5 times the upper limit of the normal reference, or estimated glomerular filtration rate (eGFR) < 45 ml/min/1.73㎡),
4. History of malignant tumors,
5. Received strong anti-osteoporosis medications such as bisphosphonates, denosumab, or teriparatide within the past 2 years,
6. History of pancreatitis or triglyceride levels >5.6 mmol/L;
7. Family history of medullary carcinoma.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
lumbar bone mineral density | From enrollment to the end of treatment at 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Xiamen University, Xiamen, Fujian, China